CLINICAL TRIAL: NCT02508337
Title: A Multicenter, Randomized, Double-masked, Vehicle-controlled, Parallel Group Phase III Study of the Efficacy and Safety of a Single Sub-conjunctival Injection of XG-102 for the Reduction of Post-cataract Surgery Intraocular Inflammation
Brief Title: Efficacy and Safety of XG-102 in Reduction of Post-cataract Surgery Intraocular Inflammation and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xigen SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDD-1002-065
Record Dates: First submitted 2015-07-20; First posted 2015-07-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Inflammation; Pain; Cataract
MeSH Terms: conditions — Inflammation; Pain; Cataract | interventions — D-JNKI-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XG-102 (Experimental): sterile ophthalmic solution for sub-conjunctival injection
  Interventions: Drug: XG-102
- placebo (Placebo Comparator): sterile ophthalmic solution for sub-conjunctival injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XG-102 — Comparison of XG-102 versus placebo for the treatment of ocular inflammation and pain associated with cataract surgery
  Arms: XG-102
Drug: Placebo — Comparison of XG-102 versus placebo for the treatment of ocular inflammation and pain associated with cataract surgery
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of XG-102 (900µg) compared to vehicle in the treatment of subjects with inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent, approved by the appropriate institutional review board;
* Be greater than or equal to 18 years of age of either sex or any race;
* Be planning to undergo unilateral cataract extraction via phacoemulsification and posterior chamber intraocular lens (PCIOL) implantation in the study eye;
* Have a pin-hole visual acuity (VA) < 1.0 logarithm of the minimum angle of resolution (logMAR) in the operative eye and fellow eye as measured using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart at Visit 1;
* (For females of childbearing potential) agree to have urine pregnancy testing performed at Visit 1 (must be negative) and at exit visit; must not be lactating; and must agree to use a medically acceptable form of birth control1 throughout the study duration. Women of childbearing potential include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).

Exclusion Criteria:

* Have a known sensitivity or allergy to the class of medication of the active ingredient in the study medication or any of the study medication's components;
* Have any intraocular inflammation (e.g., white blood cells or flare) present in the study eye at the Visit 1slit lamp examination;
* Have a score greater than "0" on the Ocular Pain Assessment at Visit 1 or 2 in the study eye;
* Have an immunosuppressive or an autoimmune disease that in the opinion of the Investigator could affect intraocular inflammation or the normal healing process of the eye;
* Have active or chronic/recurrent ocular or systemic disease that is uncontrolled and will likely affect wound healing;
* Currently have suspected or known malignancy or be currently receiving antineoplastic therapy;
* Be a female who is currently pregnant, planning a pregnancy, lactating, not using a medically acceptable form of birth control throughout the study duration, or have a positive urine pregnancy test at Visit 1;
* Use anti-inflammatory agents, analgesics/pain relievers (including opioids, narcotics and other pain medications) or immunomodulating agents, systemically, or in either eye, and/or use medications for benign prostatic hyperplasia (BPH), from the washout period through the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Absence of anterior chamber cells | Day 15
Pain scores as measured by the visual analog scale | Day2

SECONDARY OUTCOMES:
Use of rescue medication | up to D22
Number of patients with adverse events | up to D22

CONTACTS AND LOCATIONS:
Overall Officials: Juli Chalifour, Study Director — ORA, Inc.
Locations (1):
- Ora, Andover, Massachusetts, United States